CLINICAL TRIAL: NCT03950843
Title: A Multi-center, Randomized, Double-blind, Placebo Control, Therapeutic Confirmatory, Phase III Trial to Evaluate the Efficacy and Safety of CKD-825 in Patients With Atrial Fibrillation
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of CKD-825 in Patients With Atrial Fibrillation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 125AF18022
Record Dates: First submitted 2019-04-29; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): * Patients assigned to this group are treated with 1 capsule of CKD-825 and 2 placebo capsules(the placebo of CKD-825)
  * The necessity of a dose titration is adjudicated every 2 weeks.
  * After unblinding at the end of Administration Period, only patients in experimental group are treated with 1 capsule of CKD-825 for additional 4 weeks of Extension Period.
  Interventions: Drug: CKD-825; Drug: Placebo oral capsule
- Placebo Group (Placebo Comparator): * Patients assigned to this group are treated with 3 placebo capsules (the placebo of CKD-825)
  * The necessity of a dose titration is adjudicated every 2 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: CKD-825 — * Dosage Form: capsule
  * Dosage: 3 types(low/medium/high dose)
  * Frequency: QD(once daily) administration
  Other Names: Test
  Arms: Experimental Group
Drug: Placebo oral capsule — Placebo of CKD-825
  * Dosage Form: capsule
  * Dosage: NA
  * Frequency: QD administration
  Other Names: Reference

SUMMARY:
to Evaluate the Efficacy and Safety of CKD-825 in Patients With Atrial Fibrillation

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-blind, Placebo control, Therapeutic Confirmatory, Phase III Trial to Evaluate the Efficacy and Safety of CKD-825 in Patients With Atrial Fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged ≥ 19 years with persistent or permanent Atrial Fibrillation
* Patients with modified EHRA(The European Heart Rhythm Association score of atrial fibrillation) score ≥ 2a
* Patients with resting HR ≥ 80 beats per minute(bpm)
* Patients with 24-h mHR ≥ 80 bpm on Holter ECG

Exclusion Criteria:

* Treatment with antiarrhythmics within 2 weeks(Those who had washout period can be included)
* Pacemaker or implantable cardioverter defibrillator
* Catheter ablation for atrial fibrillation within 12 weeks before first investigational product(IP) administration
* Treatment for heart failure (New York Heart Association functional class 4)
* Myocardial infarction or unstable angina pectoris within 12 weeks before first IP administration
* Wolff-Parkinson-White syndrome
* Hepatic or renal disorder
* Systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg
* Uncontrolled Diabetes(HbA1c > 9%)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean 24-hour heart rate(24-h mHR) compared with the baseline value | at week 6 after first drug administration
  To compare experimental group with placebo group

SECONDARY OUTCOMES:
Change in resting heart rate(HR) on 12-lead electrocardiogram(ECG) compared with the baseline value | at week 2, week 4, week 6 and week 10 after first drug administration
  To compare experimental group with placebo group
Percentages of patients whose resting HR on 12-lead ECG achieved below 110 bpm at week 6 and week 10 among those with resting HR ≥ 110 bpm from baseline | 2 weeks, 4 weeks and 6 weeks and 10 weeks after first drug administration
  To compare experimental group with placebo group
Percentages of patients whose resting HR on 12-lead ECG achieved < 80 bpm | at week 6 and week 10 after first drug administration
  To compare experimental group with placebo group
Change in modified EHRA score(European Heart Rhythm Association score of atrial fibrillation) compared with the baseline value | at week 2, week 4, week 6 and week 10 after first drug administration
  To compare experimental group with placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Yaemin Park, M.D, Ph.D, Principal Investigator — Gachon University Gil Medical Center; Yongseog Oh, M.D, Ph.D, Principal Investigator — The Catholic University of Korea; JinBae Kim, M.D, Ph.D, Principal Investigator — Kyunghee University Hospital; Seongwook Han, M.D, Ph.D, Principal Investigator — Keimyung Universtiy Dongsan Medical Center; Jongsung Park, M.D, Ph.D, Principal Investigator — Dong-A University; Yeonggeun On, M.D, Ph.D, Principal Investigator — Samsung Medical Center; Kee-Jun Choi, M.D, Ph.D, Principal Investigator — Asan Medical Center; Sang-Weon Park, M.D, Ph.D, Principal Investigator — Sejong General Hospital; Gyo-Seung Hwang, M.D, Ph.D, Principal Investigator — Ajou University; Moon Hyoung Lee, M.D, Ph.D, Principal Investigator — Severance Hospital; Dong-Gu Shin, M.D, Ph.D, Principal Investigator — Dong-A University Hospital; Nam-Ho Kim, M.D, Ph.D, Principal Investigator — Wonkwang University Hospital; Dae-Kyeong Jun, M.D, Ph.D, Principal Investigator — Inje University; Jun Namgung, M.D, Ph.D, Principal Investigator — Inje University; Daehyeok Kim, M.D, Ph.D, Principal Investigator — Inha University Hospital; Hyung Wook Park, M.D, Ph.D, Principal Investigator — Chonnam National University Hospital; Daein Lee, M.D, Ph.D, Principal Investigator — Chugbuk National University Hospital; Hwan-Cheol Park, M.D, Ph.D, Principal Investigator — Hanyang University; Eue-Keun Choi, M.D, Ph.D, Principal Investigator — Seoul National University; Kyung Suk Lee, M.D, Ph.D, Principal Investigator — Chonbuk National University Hospital; Seon-a Jin, M.D, Ph.D, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Jong-ll, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No